CLINICAL TRIAL: NCT04204031
Title: Objective Evaluation of the Number of Use Hour of Oxygen Therapy in Patients Receiving Supplemental Oxygen
Acronym: MONOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University Hospital, Geneva (Other); Ligue Pulmonaire Genevoise (Other)
Responsible Party: Principal Investigator, Olivier Contal, Ordinary Professor HES, Haute Ecole de Santé Vaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01954
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Chronic Respiratory Failure With Hypoxia; Chronic Obstructive Pulmonary Disease
Keywords: Long term oxygen therapy; adherence; electronic monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presentation of the adherence record (Other): Following a first observation period of 15 days, participants whose actual time of use will be less than prescribed will be offered an intervention which will consist of a presentation of the adherence record. The participant will also be asked about the presence of possible barriers concerning the use of oxygen therapy. The collaborator in charge of home visits will attempt to resolve these barriers as much as possible.
  Only participants with an actual time of use less than prescribed will be offered this intervention and will continue the monitoring over a period of 15 additional days.
  Interventions: Behavioral: Presentation of the adherence record

INTERVENTIONS:
Behavioral: Presentation of the adherence record — Adherence record will be presented to participants with an actual time of use less than prescribed. The participant will also be asked about the presence of possible barriers concerning the use of oxygen therapy. The collaborator in charge of home visits will attempt to resolve these barriers as much as possible.

SUMMARY:
The aim of this study is to measure the actual use time in patients receiving supplemental oxygen using a new easy-to-use electronic remote monitoring device (TeleOx™)

DETAILED DESCRIPTION:
The first phase of the study is observational. Oxygen use time of patients with chronic respiratory failure under long term oxygen therapy will be objectively measured using a electronic remote monitoring device (TeleOx™) over 15 days. The actual use time will be compared to their oxygen prescription.

Participants whose actual time of use will be less than prescribed will be offered an intervention which will consist of a presentation of the adherence record. The participant will also be asked about the presence of possible barriers concerning the use of oxygen therapy. The collaborator in charge of home visits will attempt to resolve these barriers as much as possible. Only participants with an actual time of use less than prescribed will be offered this intervention and will continue the monitoring over a period of 15 additional days.

ELIGIBILITY:
Inclusion Criteria:

* Long term oxygeno-therapy patients in stable condition without pulmonary exacerbation in the month before inclusion
* Oxygen prescription for at least 15 hours/day

Exclusion Criteria:

* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-02 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Oxygen use time | 15 days
  Average oxygen use time (hours/day) measured with a TeleOx device

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Contal, PhD, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- Haute Ecole de Santé Vaud (HESAV), Lausanne, Switzerland